CLINICAL TRIAL: NCT02998658
Title: Barbed Versus Conventional Sutures for Vaginal Cuff Closure During Total Laparoscopic Hysterectomy. A Randomized Controlled Trial
Brief Title: Barbed Versus Conventional Sutures for Vaginal Cuff Closure During Total Laparoscopic Hysterectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Usama M Fouda, Prof., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Barbed/vaginal cuff
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Hysterectomy
Keywords: Laparoscopy; Barbed sutures; Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaginal cuff closure using barbed sutures (Experimental): Vaginal cuff is closed with barbed sutures
  Interventions: Device: Vaginal cuff closure using barbed sutures
- Vaginal cuff closure using conventional sutures (Active Comparator): Vaginal cuff is closed with conventional sutures
  Interventions: Device: Vaginal cuff closure using conventional sutures

INTERVENTIONS:
Device: Vaginal cuff closure using barbed sutures — Vaginal cuff will be closed using a 24-cm × 24-cm 0 polydioxanone double-armed suture on a 26-mm half-circle reverse cutting needle( STRATAFIX™ Spiral PDO Knotless Tissue Control Device, Ethicon Inc , Somerville, NJ, USA )
  Arms: Vaginal cuff closure using barbed sutures
Device: Vaginal cuff closure using conventional sutures — Vaginal cuff will be closed using 1-0 polyglactin 910 suture(VICRYL™.; Ethicon Inc, Sommerville, NJ) .
  Arms: Vaginal cuff closure using conventional sutures

SUMMARY:
The aim of this study is to estimate whether the use of the barbed suture facilitates laparoscopic suturing of the vaginal cuff during total laparoscopic hysterectomy.

DETAILED DESCRIPTION:
Vaginal cuff suturing is a significant step during hysterectomy with regard to operating time and a critical passage for the risk of vaginal cuff dehiscence. Vaginal cuff dehiscence is a severe adverse event and occurs more frequently after total laparoscopic hysterectomy (0.3-3.1 %) compared to abdominal and vaginal hysterectomy

Barbed suture is a new type of sutures introduced to facilitate laparoscopic suturing.When compared with conventional smooth suture, barbed suture has external barbs that anchor the suture to the tissues and prevent the retrograde movement of suture thread during suturing. Consequently, laparoscopic suturing can be performed easily without the need for suture locking, without applying traction on suture thread by the assistant and without tying knots at both ends of the suture line In gynecology, barbed sutures have been used in minimally invasive ,myomectomy hysterectomy, ovarian cystectomy and sacrocolpopexy. There is a growing body of evidence that the use of barbed sutures in these procedures facilitates laparoscopic suturing and significantly reduces suturing time, total operating time and intraoperative blood loss To date only two small randomized controlled trials compared the effectiveness of the bidirectional knotless barbed suture versus standard suture in the repair of vaginal cuff

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication for hysterectomy ( i.e. pain, bleeding and pressure symptoms)

Exclusion Criteria:

* Genital malignancy
* Uterine size more than 16 weeks
* Coagulation defects or concurrent anticoagulant therapy
* Pregnancy
* Compromised cardiopulmonary status
* Contraindications for general anesthesia

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2017-02; Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Suturing time of vaginal cuff | During hysterectomy operation

SECONDARY OUTCOMES:
Operative time | During hysterectomy operation

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, Prof., Study Director — Cairo university ,Faculty of medicine , Obstetrics and Gynecology Department; Khaled A Elsetohy,, Prof., Principal Investigator — Cairo university ,Faculty of medicine , Obstetrics and Gynecology Department
Locations (1):
- Cairo university, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Einarsson JI, Cohen SL, Gobern JM, Sandberg EM, Hill-Lydecker CI, Wang K, Brown DN. Barbed versus standard suture: a randomized trial for laparoscopic vaginal cuff closure. J Minim Invasive Gynecol. 2013 Jul-Aug;20(4):492-8. doi: 10.1016/j.jmig.2013.02.015. Epub 2013 May 14. PMID 23680517